CLINICAL TRIAL: NCT07222462
Title: ASTRAL: A Superiority Trial of Radiofrequency Ablation for Low Back Pain
Brief Title: A Superiority Trial of Radiofrequency Ablation for Low Back Pain
Acronym: ASTRAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Janna Friedly, Multiple Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00075903; U01AR084723 (NIH)
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: lumbar radiofrequency ablation (LRFA); corticosteroid injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LRFA-C (Active Comparator): Lumbar radiofrequency ablation with conventional electrodes
  Interventions: Procedure: Lumbar radiofrequency ablation with conventional electrodes (LRFA-C)
- LRFA-M (Active Comparator): Lumbar radiofrequency ablation with multi-tined electrodes
  Interventions: Procedure: Lumbar radiofrequency ablation with multi-tined electrodes (LRFA-M)
- Simulated LRFA (Sham Comparator): Simulated lumbar radiofrequency ablation
  Interventions: Procedure: Simulated lumbar radiofrequency ablation

INTERVENTIONS:
Procedure: Lumbar radiofrequency ablation with conventional electrodes (LRFA-C) — LRFA-C positions a conventional thermal radiofrequency electrode at each medial branch nerve to be ablated and administers local anesthetic to the nerve. Parallel placement of the electrode will be achieved. Once the electrode is in correct position and nerve stimulation testing done, a radiofrequency lesion is generated, achieving a temperature 80°C-90°C, lasting 90-120 seconds. If a 16-gauge or larger electrode is used, no second lesion needs to be made. If an 18-gauge electrode is used, the electrode will be repositioned slightly by withdrawing or repositioning parallel to the 1st ablation site, or by rotating the electrode, and a 2nd lesion made. Local corticosteroid injection is then performed at the ablation site at a total corticosteroid equivalent of 80mg triamcinolone, divided equally among the medial branches targeted; this dose can be reduced as needed according to the medical status of each patient. This process is applied for each medial branch nerve targeted.
  Arms: LRFA-C
Procedure: Lumbar radiofrequency ablation with multi-tined electrodes (LRFA-M) — LRFA-M positions a multi-tined thermal radiofrequency electrode at each medial branch nerve to be ablated and administers local anesthetic to the nerve. However, the multi-tined thermal radiofrequency electrode is thought to achieve larger lesions and thus does not require parallel electrode placement; the LRFA-M electrode will be placed perpendicular to the medial branch nerve. All subsequent processes are the same as for LRFA-C. This includes local corticosteroid injection at each ablation site at a total corticosteroid equivalent of 80mg triamcinolone, divided equally among the medial branches targeted; this dose can be reduced as needed according to the medical status of each patient. This process is applied for each medial branch nerve targeted.
  Arms: LRFA-M
Procedure: Simulated lumbar radiofrequency ablation — The simulated LRFA control procedure will be performed in an identical fashion to LRFA-M, except 1) after electrode positioning, a neurodestructive lesion will not be made; and 2) a pre-recorded audio recording of the procedure will be played (out of view of the patient, immediately adjacent to the RFA machine) in order to simulate the beeping and other sounds of the machine and to ensure the appropriate length of the simulated procedure. The electrode will remain in place for the 90-120 seconds that lesioning would normally take, but without heat application. The electrode will then be repositioned to simulate a second lesion, also of duration 90-120 seconds. Local corticosteroid injection is then performed at the ablation site at a total corticosteroid equivalent of 80mg triamcinolone, divided equally among the medial branches targeted; this dose can be reduced as needed according to the medical status of each patient. This process is applied for each medial branch nerve targeted.
  Arms: Simulated LRFA

SUMMARY:
The purpose of the ASTRAL Study is to evaluate the effectiveness of LRFA (Lumbar radiofrequency ablation) against a control procedure. The ASTRAL Study will enroll individuals with chronic low back pain (CLBP) and randomly assign them to one of three groups: lumbar radiofrequency ablation using conventional electrodes placed parallel to the medial branch nerves (LRFA-C), lumbar radiofrequency ablation using multi-tined electrodes placed perpendicular to the medial branch nerves (LRFA-M), or a simulated radiofrequency ablation procedure.

DETAILED DESCRIPTION:
Low back pain is the #1 contributor to years lived with disability in the United States. Lumbar radiofrequency ablation (LRFA) is a minimally invasive procedure for chronic low back pain (CLBP) commonly used in the US, but the effectiveness of this procedure has yet to be fully explored, and a definitive, double-blind, multicenter RCT demonstrating a clinically relevant benefit of LRFA over a control procedure has yet to be conducted. LRFA-C involves placing a conventional radiofrequency electrode parallel to each targeted medial branch nerve, administering local anesthetic, and confirming placement with nerve stimulation as per standard clinical practice. LRFA-M follows the same processes as LRFA-C, albeit a multi-tined radiofrequency electrode will be used to create larger lesions, and the electrode will be positioned perpendicular to the medial branch nerve. The primary objectives of ASTRAL are to 1) compare the effectiveness of LRFA-C with a simulated LRFA control procedure for improving back-related functional limitations, and 2) compare the effectiveness of LRFA-M with a simulated LRFA control procedure for improving back-related functional limitations. The ASTRAL Study also aims to explore the difference in effectiveness, procedure duration, radiation dosage, and pain intensity between LRFA-C and LRFA-M.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* CLBP of duration ≥ 3 months. Low back pain is defined as occurring between the lower posterior margin of the rib cage and the horizontal gluteal fold.
* Low back pain intensity numerical rating scale (NRS) ≥ 4 with one of the following prior to LRFA: 1) Current low back pain intensity, 2) Average pain over past 7 days, OR 3) Pain intensity without specification of recall period
* Has had conservative treatments for CLBP (physical therapy, exercise therapy, spinal manipulation, massage, acupuncture, etc.)
* Candidate for unilateral LRFA (L1-S1 joints; ≤3 levels); or bilateral LRFA (L1-S1 joints; ≤2 levels)
* 'Positive responses' (≥80% improvement of CLBP pain intensity) to 2 sets of anesthetic-only MBBs (≤0.5cc of local anesthetic)
* Able to read, speak, and understand English sufficient for informed consent purposes
* Stated willingness to comply with all study processes and availability for the duration of the study, and provision of a signed and dated informed consent form

Exclusion Criteria:

* CLBP attributed primarily to specific spine-related conditions (radiculopathy, lumbar spinal stenosis, spinal instability), 'red flag' conditions (infection / malignancy / fracture), and/or inflammatory arthritis (RA, SpA, etc.)
* Prior LRFA
* Prior lumbar facet joint (intra-articular or medial branch nerve) corticosteroid injections (past 6 months)
* Surgery involving one or more of spinal levels where LRFA is to be performed, in the past 2 years
* Lumbar fusion involving the spinal levels where LRFA is considered, at any time
* Prior known severe lumbar central canal stenosis on MRI as defined by Lee (2011): obliteration of the cerebrospinal fluid (CSF), and marked compression of dural sac, and none of the cauda equina can be visually separated from each other. No new MRIs would be done specifically as part of the study processes.
* Prior formal diagnosis of fibromyalgia by a rheumatologist (diagnosis by primary care physician or pain medicine specialist is not sufficient)
* Unstable psychiatric or terminal medical conditions that would limit study participation and the likelihood of follow-up for 12 months post-randomization
* Pregnancy, being a prisoner, or having a prior formal diagnosis of cognitive impairment by a neuropsychologist or neurologist, confirmed by health record documentation
* Participant report of prior formal diagnosis of cognitive impairment by a neuropsychologist or neurologist can be obtained, but participant-reported cognitive impairment by a neuropsychologist or neurologist must be confirmed via health record documentation. No new evaluations for cognitive impairment would be done specifically as part of the study processes.
* Contraindication to local anesthetic, corticosteroid, or any aspects of LRFA
* Cannot reach MBB targets with 11.9cm needle
* Major planned life events over the next 4 months that might interfere with study participation (e.g., major abdominal or chest surgery or extended vacation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Back-related functional limitations | 3 months post-randomization
  Measured using the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that evaluates patients' self-reported functional limitations due to back pain. The total score ranges from 0 (no disability) to 24 (severe disability).

SECONDARY OUTCOMES:
Back-related functional limitations | 1 month post-randomization
  Measured using the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that evaluates patients' self-reported functional limitations due to back pain. The total score ranges from 0 (no disability) to 24 (severe disability).
Back-related functional limitations | 6 months post-randomization
  Measured using the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that evaluates patients' self-reported functional limitations due to back pain. The total score ranges from 0 (no disability) to 24 (severe disability).
Back-related functional limitations | 12 months post-randomization
  Measured using the Roland-Morris Disability Questionnaire (RMDQ), a 24-item questionnaire that evaluates patients' self-reported functional limitations due to back pain. The total score ranges from 0 (no disability) to 24 (severe disability).
Procedure duration | Day of intervention, after procedure
  Duration of the procedure in minutes
Radiation dose | Day of intervention, after procedure
  Total radiation used during procedure
Participant pain during the procedure | Day of intervention, after procedure
  Patient low back pain intensity experienced during the procedure will be assessed within 1 hour after the procedure, using the average of (a) patient rating of average pain intensity as experienced during the procedure and (b) patient rating of worst pain intensity as experienced during the procedure. The scale for each of these two items ranges from 0 (no pain) to 10 (worst pain imaginable).
Pain intensity | 3 months post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain intensity item, asking about low back pain specifically. The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain intensity | 1 month post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain intensity item, asking about low back pain specifically. The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain intensity | 6 months post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain intensity item, asking about low back pain specifically. The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain intensity | 12 months post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain intensity item, asking about low back pain specifically. The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain interference | 3 months post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain interference item, asking about interference due to low back pain specifically. The scale ranges from 0 (no interference) to 10 (complete interference).
Pain interference | 1 month post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain interference item, asking about interference due to low back pain specifically. The scale ranges from 0 (no interference) to 10 (complete interference).
Pain interference | 6 months post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain interference item, asking about interference due to low back pain specifically. The scale ranges from 0 (no interference) to 10 (complete interference).
Pain interference | 12 months post-randomization
  Measured using the Pain, Enjoyment of Life, and General Activity (PEG) Scale pain interference item, asking about interference due to low back pain specifically. The scale ranges from 0 (no interference) to 10 (complete interference).
Time to receiving other procedural treatment for CLBP | 12 months post-randomization
  From post-randomization, the number of days to receiving any other procedural treatment for CLBP

OTHER OUTCOMES:
Quality of life (EuroQoL 5-item) | 3 months post-randomization
  Measured using the EuroQoL 5 Dimension (EQ-5D). The first component of the EuroQoL contains 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each of which has three response levels. These items produce a 0 to 1 score, with higher scores indicating better health.
Quality of life (EuroQoL 5-item) | 1 month post-randomization
  Measured using the EuroQoL 5 Dimension (EQ-5D). The first component of the EuroQoL contains 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each of which has three response levels. These items produce a 0 to 1 score, with higher scores indicating better health.
Quality of life (EuroQoL 5-item) | 6 months post-randomization
  Measured using the EuroQoL 5 Dimension (EQ-5D). The first component of the EuroQoL contains 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each of which has three response levels. These items produce a 0 to 1 score, with higher scores indicating better health.
Quality of life (EuroQoL 5-item) | 12 months post-randomization
  Measured using the EuroQoL 5 Dimension (EQ-5D). The first component of the EuroQoL contains 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each of which has three response levels. These items produce a 0 to 1 score, with higher scores indicating better health.
Quality of life (VAS) | 3 months post-randomization
  The second component of the EuroQOL is a visual analog scale asking participants to rate their health from 0-100, with higher ratings indicating better health.
Quality of life (VAS) | 1 month post-randomization
  The second component of the EuroQOL is a visual analog scale asking participants to rate their health from 0-100, with higher ratings indicating better health.
Quality of life (VAS) | 6 months post-randomization
  The second component of the EuroQOL is a visual analog scale asking participants to rate their health from 0-100, with higher ratings indicating better health.
Quality of life (VAS) | 12 months post-randomization
  The second component of the EuroQOL is a visual analog scale asking participants to rate their health from 0-100, with higher ratings indicating better health.
Physical functioning | 3 months post-randomization
  Measured using the PROMIS Physical Functioning SF-6B, consisting of 6 questions regarding abilities for daily functions and activities. Scores range from 0 to 100, with higher scores indicating greater function. Scores are normalized to a mean of 50 and standard deviation of 10.
Physical functioning | 1 month post-randomization
  Measured using the PROMIS Physical Functioning SF-6B, consisting of 6 questions regarding abilities for daily functions and activities. Scores range from 0 to 100, with higher scores indicating greater function. Scores are normalized to a mean of 50 and standard deviation of 10.
Physical functioning | 6 months post-randomization
  Measured using the PROMIS Physical Functioning SF-6B, consisting of 6 questions regarding abilities for daily functions and activities. Scores range from 0 to 100, with higher scores indicating greater function. Scores are normalized to a mean of 50 and standard deviation of 10.
Physical functioning | 12 months post-randomization
  Measured using the PROMIS Physical Functioning SF-6B, consisting of 6 questions regarding abilities for daily functions and activities. Scores range from 0 to 100, with higher scores indicating greater function. Scores are normalized to a mean of 50 and standard deviation of 10.
Depression | 3 months post-randomization
  Measured using the Patient Health Questionnaire (PHQ-2), consisting of 2 questions regarding frequency of depressive symptoms on a level from 0 (not at all) to 3 (nearly every day).
Depression | 1 month post-randomization
  Measured using the Patient Health Questionnaire (PHQ-2), consisting of 2 questions regarding frequency of depressive symptoms on a level from 0 (not at all) to 3 (nearly every day).
Depression | 6 months post-randomization
  Measured using the Patient Health Questionnaire (PHQ-2), consisting of 2 questions regarding frequency of depressive symptoms on a level from 0 (not at all) to 3 (nearly every day).
Depression | 12 months post-randomization
  Measured using the Patient Health Questionnaire (PHQ-2), consisting of 2 questions regarding frequency of depressive symptoms on a level from 0 (not at all) to 3 (nearly every day).
Anxiety | 3 months post-randomization
  Measured using the Generalized Anxiety Disorder Scale (GAD-2), consisting of 2 questions regarding frequency of anxiety on a level from 0 (not at all) to 3 (nearly every day).
Anxiety | 1 month post-randomization
  Measured using the Generalized Anxiety Disorder Scale (GAD-2), consisting of 2 questions regarding frequency of anxiety on a level from 0 (not at all) to 3 (nearly every day).
Anxiety | 6 months post-randomization
  Measured using the Generalized Anxiety Disorder Scale (GAD-2), consisting of 2 questions regarding frequency of anxiety on a level from 0 (not at all) to 3 (nearly every day).
Anxiety | 12 months post-randomization
  Measured using the Generalized Anxiety Disorder Scale (GAD-2), consisting of 2 questions regarding frequency of anxiety on a level from 0 (not at all) to 3 (nearly every day).
Pain catastrophizing | 1 month post-randomization
  Measured using the Pain Catastrophizing Scale (PCS) SF-6, consisting of 6 questions regarding frequency of pain catastrophizing on a level from 0 (not at all) to 4 (all the time).
Pain catastrophizing | 3 months post-randomization
  Measured using the Pain Catastrophizing Scale (PCS) SF-6, consisting of 6 questions regarding frequency of pain catastrophizing on a level from 0 (not at all) to 4 (all the time).
Pain catastrophizing | 6 months post-randomization
  Measured using the Pain Catastrophizing Scale (PCS) SF-6, consisting of 6 questions regarding frequency of pain catastrophizing on a level from 0 (not at all) to 4 (all the time).
Pain catastrophizing | 12 months post-randomization
  Measured using the Pain Catastrophizing Scale (PCS) SF-6, consisting of 6 questions regarding frequency of pain catastrophizing on a level from 0 (not at all) to 4 (all the time).
Substance use (tobacco) | 3 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The tobacco item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (tobacco) | 1 month post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The tobacco item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (tobacco) | 6 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The tobacco item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (tobacco) | 12 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The tobacco item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (alcohol) | 3 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The alcohol item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (alcohol) | 1 month post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The alcohol item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (alcohol) | 6 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The alcohol item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (alcohol) | 12 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The alcohol item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (prescription drugs) | 3 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The prescription drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (prescription drugs) | 1 month post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The prescription drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (prescription drugs) | 6 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The prescription drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (prescription drugs) | 12 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The prescription drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (drugs) | 3 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (drugs) | 1 month post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (drugs) | 6 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Substance use (drugs) | 12 months post-randomization
  Measured using the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS-1) Tool, consisting of 4 multiple choice questions regarding frequency of substance use in the last 12 months. Each item is rated on a 5-point Likert scale from 0 (daily to almost daily) to 4 (never). The drugs item will be evaluated as a separate outcome, where any score above 0 indicates having a positive screen.
Global impression of change | 3 months post-randomization
  Measured using the Patient Global Impression of Change (PGIC) scale, ranging from 1 (no change or worse) to 7 (a great deal better).
Global impression of change | 1 month post-randomization
  Measured using the Patient Global Impression of Change (PGIC) scale, ranging from 1 (no change or worse) to 7 (a great deal better).
Global impression of change | 6 months post-randomization
  Measured using the Patient Global Impression of Change (PGIC) scale, ranging from 1 (no change or worse) to 7 (a great deal better).
Global impression of change | 12 months post-randomization
  Measured using the Patient Global Impression of Change (PGIC) scale, ranging from 1 (no change or worse) to 7 (a great deal better).
Sleep disturbance | 3 months post-randomization
  Measured using the PROMIS Sleep Disturbance SF-6A, consisting of 6 multiple choice questions (each containing five levels) regarding quality of sleep. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Sleep disturbance | 1 month post-randomization
  Measured using the PROMIS Sleep Disturbance SF-6A, consisting of 6 multiple choice questions (each containing five levels) regarding quality of sleep. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Sleep disturbance | 6 months post-randomization
  Measured using the PROMIS Sleep Disturbance SF-6A, consisting of 6 multiple choice questions (each containing five levels) regarding quality of sleep. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Sleep disturbance | 12 months post-randomization
  Measured using the PROMIS Sleep Disturbance SF-6A, consisting of 6 multiple choice questions (each containing five levels) regarding quality of sleep. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Sleep duration | 3 months post-randomization
  Measured using a self-reported measure of average nightly hours of sleep from the past month.
Sleep duration | 1 month post-randomization
  Measured using a self-reported measure of average nightly hours of sleep from the past month.
Sleep duration | 6 months post-randomization
  Measured using a self-reported measure of average nightly hours of sleep from the past month.
Sleep duration | 12 months post-randomization
  Measured using a self-reported measure of average nightly hours of sleep from the past month.
Opioid use | 3 months post-randomization
  Measured using the self-reported Morphine-Equivalent Daily Dose (MED), a measure that assesses frequency and dosage of opioids.
Opioid use | 1 month post-randomization
  Measured using the self-reported Morphine-Equivalent Daily Dose (MED), a measure that assesses frequency and dosage of opioids.
Opioid use | 6 months post-randomization
  Measured using the self-reported Morphine-Equivalent Daily Dose (MED), a measure that assesses frequency and dosage of opioids.
Opioid use | 12 months post-randomization
  Measured using the self-reported Morphine-Equivalent Daily Dose (MED), a measure that assesses frequency and dosage of opioids.
Patient prioritized functional limitations and activities | 3 months post-randomization
  Measured using the Patient-Specific Functional Scale, consisting of 5 items that ask the patient to report activities they have difficulty completing due to their low back pain, rating the difficulty level of each activity from 1 (unable to complete) to 10 (able to perform at same level as before).
Patient prioritized functional limitations and activities | 1 month post-randomization
  Measured using the Patient-Specific Functional Scale, consisting of 5 items that ask the patient to report activities they have difficulty completing due to their low back pain, rating the difficulty level of each activity from 1 (unable to complete) to 10 (able to perform at same level as before).
Patient prioritized functional limitations and activities | 6 months post-randomization
  Measured using the Patient-Specific Functional Scale, consisting of 5 items that ask the patient to report activities they have difficulty completing due to their low back pain, rating the difficulty level of each activity from 1 (unable to complete) to 10 (able to perform at same level as before).
Patient prioritized functional limitations and activities | 12 months post-randomization
  Measured using the Patient-Specific Functional Scale, consisting of 5 items that ask the patient to report activities they have difficulty completing due to their low back pain, rating the difficulty level of each activity from 1 (unable to complete) to 10 (able to perform at same level as before).
Pain frequency (P-FIBS) | 3 months post-randomization
  Measured using the Pain Frequency, Intensity, and Burden Scale (P-FIBS), consisting of 4 questions rating the frequency of pain from 0 (never) to 8 (every day).
Pain frequency (P-FIBS) | 1 month post-randomization
  Measured using the Pain Frequency, Intensity, and Burden Scale (P-FIBS), consisting of 4 questions rating the frequency of pain from 0 (never) to 8 (every day).
Pain frequency (P-FIBS) | 6 months post-randomization
  Measured using the Pain Frequency, Intensity, and Burden Scale (P-FIBS), consisting of 4 questions rating the frequency of pain from 0 (never) to 8 (every day).
Pain frequency (P-FIBS) | 12 months post-randomization
  Measured using the Pain Frequency, Intensity, and Burden Scale (P-FIBS), consisting of 4 questions rating the frequency of pain from 0 (never) to 8 (every day).
Pain frequency (ordinal) | 3 months post-randomization
  Measured using the NIH Minimal Dataset (MDS) pain frequency item that measures frequency of back pain in the past 6 months, where higher scores represent more frequent pain.
Pain frequency (ordinal) | 1 month post-randomization
  Measured using the NIH Minimal Dataset (MDS) pain frequency item that measures frequency of back pain in the past 6 months, where higher scores represent more frequent pain.
Pain frequency (ordinal) | 6 months post-randomization
  Measured using the NIH Minimal Dataset (MDS) pain frequency item that measures frequency of back pain in the past 6 months, where higher scores represent more frequent pain.
Pain frequency (ordinal) | 12 months post-randomization
  Measured using the NIH Minimal Dataset (MDS) pain frequency item that measures frequency of back pain in the past 6 months, where higher scores represent more frequent pain.
Concurrent analgesic use | 3 months post-randomization
  Measured using a self-report item inquiring about pain medications (any) used in the past 24 hours. This is a binary variable (any use vs. no use in past 24 hours).
Concurrent analgesic use | 1 month post-randomization
  Measured using a self-report item inquiring about pain medications (any) used in the past 24 hours. This is a binary variable (any use vs. no use in past 24 hours).
Concurrent analgesic use | 6 months post-randomization
  Measured using a self-report item inquiring about pain medications (any) used in the past 24 hours. This is a binary variable (any use vs. no use in past 24 hours).
Concurrent analgesic use | 12 months post-randomization
  Measured using a self-report item inquiring about pain medications (any) used in the past 24 hours. This is a binary variable (any use vs. no use in past 24 hours).
Pain intensity after accounting for concurrent analgesic use | 3 months post-randomization
  Measured using a self-reported pain intensity without medications item on a numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain intensity after accounting for concurrent analgesic use | 1 month post-randomization
  Measured using a self-reported pain intensity without medications item on a numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain intensity after accounting for concurrent analgesic use | 6 months post-randomization
  Measured using a self-reported pain intensity without medications item on a numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Pain intensity after accounting for concurrent analgesic use | 12 months post-randomization
  Measured using a self-reported pain intensity without medications item on a numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Physical activity (moderate vs. vigorous) | 3 months post-randomization
  Measured using the Behavioral Risk Factor Surveillance System (BRFSS) Physical Activity Self-report, assessing frequency and time spent participating in vigorous and moderate activity in the past week. These values will be converted to moderate-equivalent minutes using the formula: Moderate-equivalent minutes = (Moderate minutes) + (Vigorous minutes × 2).
Physical activity (moderate vs. vigorous) | 1 month post-randomization
  Measured using the Behavioral Risk Factor Surveillance System (BRFSS) Physical Activity Self-report, assessing frequency and time spent participating in vigorous and moderate activity in the past week. These values will be converted to moderate-equivalent minutes using the formula: Moderate-equivalent minutes = (Moderate minutes) + (Vigorous minutes × 2).
Physical activity (moderate vs. vigorous) | 6 months post-randomization
  Measured using the Behavioral Risk Factor Surveillance System (BRFSS) Physical Activity Self-report, assessing frequency and time spent participating in vigorous and moderate activity in the past week. These values will be converted to moderate-equivalent minutes using the formula: Moderate-equivalent minutes = (Moderate minutes) + (Vigorous minutes × 2).
Physical activity (moderate vs. vigorous) | 12 months post-randomization
  Measured using the Behavioral Risk Factor Surveillance System (BRFSS) Physical Activity Self-report, assessing frequency and time spent participating in vigorous and moderate activity in the past week. These values will be converted to moderate-equivalent minutes using the formula: Moderate-equivalent minutes = (Moderate minutes) + (Vigorous minutes × 2).

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Suri, MD, Principal Investigator — University of Washington; Janna Friedly, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Emory Musculoskeletal Institute, Atlanta, Georgia
  - Cleveland Clinic, Cleveland, Ohio
  - University of Utah Orthopaedic Center/PM&R, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data types for the full ASTRAL sample will include patient-reported outcome data; clinical and sociodemographic data entered by participants or by research staff at the clinical research center sites (CRCs) based on electronic health record (EHR) review; and adverse event monitoring data entered by participants or by research staff at the CRCs after EHR review. These de-identified, individual level data will be made available through a data repository consistent with NIH recommendations at the time of, for sharing to approved users via CSV files.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will share a complete, cleaned, de-identified copy of the locked final dataset used in conducting the final analyses upon which the accepted primary study publication is based. Data will be made available no later than when the first manuscript reporting on 12-month outcomes is published, or end of the performance period, whichever comes first. A complete dataset will be permanently archived and available through Zenodo, a generalist repository providing long-term access to and preservation of data.
Access Criteria: Registered and approved users of the data must propose specific research questions in an analysis plan and sign a data use agreement (DUA). Documentation will be made available including the study protocol, the final data management and sharing plan, data dictionary/codebook, a statistical analysis plan, data collection instruments, informed consent document, and citations to the main publications based on analyses of data being deposited. For approved requests, data made available via Zenodo will include the de-identified analyzable dataset in CSV format, data variable and value labeling guidelines, and analytic code (including code used to create derived variables).

REFERENCES:
- See also: ASTRAL Study general information website — http://www.astralstudy.org